CLINICAL TRIAL: NCT06206395
Title: Assiut University-Egypt
Brief Title: Role of Multi-modality Imaging in the Assessment of Chemotherapy Related Cardiac Dysfunction Among Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, John Safwat Johny, Assiut University, Assiut University
Other Study IDs: Cardiotoxicity and cancer
Record Dates: First submitted 2023-09-25; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: 2D Speckle Tracking Echocardiography; Breast Cancer; Cardiac Magnetic Resonance
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients receiving chemotherapeutic drugs: Cancer patients ≥ 18 years of age, and scheduled to receive chemotherapy will be included.
  Interventions: Device: Two dimensions speckle tracking and three dimension echocardiography and cardiac magnetic resonance imaging

INTERVENTIONS:
Device: Two dimensions speckle tracking and three dimension echocardiography and cardiac magnetic resonance imaging — 2D speckle tracking echo will be performed before chemotherapy and after mid-cycle and after completion of treatment.
  3D echo and CMR will be performed before and after chemotherapy treatment.

SUMMARY:
The field of oncology has advanced remarkably. Some of the old and new emerging cancer therapies are associated with development of cardiovascular toxicities , which may have the potential to offset the gains in survival obtained with this cancer treatment advances. Much of the focus on cardiovascular toxicities has been in the early detection of myocardial damage and prediction of cancer therapeutics-related cardiac dysfunction (CTRCD). The main strategy for these patients is timely diagnosis and treatment of high-risk individual Cardiac dysfunction associated with cancer treatment is the main cause of mortality in cancer survivors. The mortality rate is recorded to be up to 60% in the first two years after therapy. The most commonly associated drugs with cardiotoxicity are anthracycline (AC) and monoclonal antibodies (such as trastuzumab). Other new agents, such as vascular endothelial growth factor (VEGF) inhibitors, immunotherapies, and proteasome inhibitors, can also cause cardiac dysfunction .

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients ≥ 18 years of age, and scheduled to receive chemotherapy will be included.

Exclusion Criteria:

* Contraindications to CMR (e.g.: patients with pacemakers, defibrillators or other implanted electronic devices).
* Life expectancy ≤ 12 months.
* Participating in another oncology clinical trial;
* Prior exposure to chemotherapy;
* History of active or prior cardiac disease (e.g., myocardial infarction, heart failure or base line left ventricular ejection fraction less than 55%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients receiving chemotherapeutic drugs with or without adjuvant radiotherapy at oncology department of Assiut University Hospital will be enrolled and imaging modalities will be performed at Assiut University Heart Hospital.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Determine and compare the role of 2D speckle tracking vs. 3D echocardiography in assessment of early LV systolic dysfunction in patients receiving different chemotherapy combinations | up to 6 months after starting chemotherapy
  All patient will be undergo both 2D and 3D echocardiography before and after treatment to detect early LV systolic dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: John S Johny, MSC, Principal Investigator — Assiut University
Locations (1):
- Assiut University-Cardiovascular department, Asyut, Egypt